CLINICAL TRIAL: NCT01131429
Title: Survival Analysis of A Chinese Randomized Crossover Study Comparing Erlotinib to Docetaxel/Cisplatin in Previously Untreated Stage IIIB/IV Lung Adenocarcinoma With EGFR Mutations
Brief Title: A Chinese Randomized Crossover Study of Erlotinib Versus Docetaxel/Cisplatin in Previously Untreated Stage IIIB/IV Lung Adenocarcinoma With EGFR Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Liang-An Chen, M.D., Ph.D, Chinese PLA General Hospital, Beijing, China
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PLAGH-TKIs
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-04

CONDITIONS: Neoplasms, Lung; Carcinoma, Non-Small Cell Lung; Drug Therapy; Genes, EGFR
Keywords: mutation analysis; first-line; second-line; targeted therapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- first-line erlotinib (Experimental): erlotinib in first-line treatment and docetaxel/cisplatin in second-line treatment
  Interventions: Drug: Erlotinib; Drug: Docetaxel; Drug: Cisplatin
- second-line erlotinib (Active Comparator): docetaxel/cisplatin in first-line treatment and erlotinib in second-line treatment
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg/d per os until proven disease progression
  Arms: first-line erlotinib
Drug: Docetaxel — Docetaxel 75mg/m2 iv day 1 every 3 weeks as second-line treatment
  Arms: first-line erlotinib
Drug: Cisplatin — cisplatin 75mg/ m2 iv day 1 every 3 weeks as second-line treatment
  Arms: first-line erlotinib
Drug: Docetaxel — Docetaxel 75mg/m2 iv day 1 every 3 weeks for 6 cycles at most
  Arms: second-line erlotinib
Drug: Cisplatin — Cisplatin 75mg/m2 iv day 1 every 3 weeks for 6 cycles at most
  Arms: second-line erlotinib
Drug: Erlotinib — Erlotinib 150 mg/d per os as second-line treatment
  Arms: second-line erlotinib

SUMMARY:
Objective: the objective of this study in china is to clarify, whether the overall survival is different between previously untreated stage IIIB/IV lung adenocarcinoma with EGFR mutations receiving first-line erlotinib plus second-line docetaxel/cisplatin and those receiving first-line docetaxel/cisplatin plus second-line erlotinib .

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged over 18 years
* Histologically proven lung adenocarcinoma
* clinical stage IIIB/IV
* ECOG performance status 0-2
* Had no prior anticancer agent, radiation or surgical therapy for lung adenocarcinoma
* At least one measurable lesion (according to RECIST)
* Provision of written informed consent
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* History of malignant disease.
* Evidence of clinically active interstitial lung diseases (patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded)
* Expected life expectancy less than 2 months
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) ≥ 2.5 x ULN if no demonstrable liver metastases (or >5 x in presence of liver metastases)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
* Pregnancy or breast-feeding women (women of child¬bearing potential). Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | three year

SECONDARY OUTCOMES:
progression-free survival during the first-line treatment | 1 year
progression-free time during the second-line treatment | 2 years
quality of life during the first-line therapy | every 3 weeks during first-line therapy
quality of life during the second-line therapy | every 3 weeks during the second-line therapy
response rates during the first-line treatment | at 6 months from treatment initiation
response rates during the second-line treatment | every 3 weeks during the treament, and and every 6 weeks thereafter
toxicity during the first-line treatment | at 12 months from treatment initiation
toxicity during the second-line treatment | end of study
preditive and prognostic markers for chemotherapy or erlotinib | end of study
  tissues for markers analysis are acquired during diagnosis procedure with informed consent.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-An Chen, M.D., Ph.D., Study Chair — Chinese PLA General Hospital, Beijing, China
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China